CLINICAL TRIAL: NCT03461562
Title: Effectiveness of Exercise Applications on Hepatic Steatosis and Physical Fitness in Patients With Nonalcholic Fatty Liver Disease
Brief Title: Effectiveness of Exercise Applications on Hepatic Steatosis and Physical Fitness in Patients With NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Marmara University (Other); Medipol University (Other)
Responsible Party: Principal Investigator, Tülay Çevik, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEDIPOL UNIVERSITY
Record Dates: First submitted 2018-02-27; First posted 2018-03-12 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Aerobic Exercise; Whole Body Vibration Therapy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Other: Aerobic Exercise
- Control (Active Comparator)
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Aerobic exercise wil be held for 40 minutes. Dynamic exercises will be accompanied by physiotherapist on the vibration platform for 15 minutes. Same excercises will be held stable platform (when the devices turned off) by control group for 15 minutes.
  Other Names: Whole Body Vibration Therapy

SUMMARY:
Purpose of the study will investigate the effects of two different training programs on hepatic steatosis and physical fitness parameters. This trial is designed in a randomized controlled study plan and aerobic training (40 minutes) wil be combined with Whole Body Vibration Training (WBVT for 15 minutes) which is made up of a shorter time application. WBVT to be applied instead of the resistance exercises.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NAFLD
* Age range of 18-65 years
* Participants who are not in an active exercise program
* Participants who are not on an active diet program

Exclusion Criteria:

* Pregnancy
* Chronic inflammatory process
* Rheumatic disease
* Cognitive disorders
* Obstacles to achieve physical performance tests
* Presence of other conditions that may cause liver steatosis
* Inability to do WBVT or Aerobic Exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
FibroScan | 8 weeks
  İn the Fibroscan measurement session, the patient lying supine, the tip of the transducer is placed on the skin between the ribs over the right lobe of the liver. At least 10 validated measurements with a ratio of interquartile range (IQR) and median LSM of less than or equal to 30 percent are required for an interpretation of significant fibrosis or cirrhosis.

SECONDARY OUTCOMES:
Profile of liver enzymes | 8 weeks
  Serum liver enzymes ALT, AST, GGT, ALP will be recorded.

OTHER OUTCOMES:
Body composition | 8 weeks
  Body mass index (BMI) will be calculated by dividing weight (kg) by height (m2).
  The BMI Categories will be done as follows:
  Underweight = <18.5 Normal weight = 18.5-24.9 Overweight = 25-29.9 Obesity = BMI of 30 or greater
Cardiopulmonary exercise testing | 8 weeks
  Cardiopulmonary exercise testing (CPET) will be done.The goal of testing is to evaluate the physiologic response of the heart, lungs and muscles to an increase in physical stress. Cardiopulmonary exercise testing (CPET) with cycle ergometer.
  The following values will be calculated personally. Peak oxygen consumption Peak heart rate Metabolic equivalent Aerobic threshold Anaerobic threshold Heart rate reserve
Body Fat Percentage | 8 weeks
  Body Fat Percentage will be calculated skinfold measures using Jackson-Pollock measurement system. The Jackson-Pollack method for evaluating body fat percentage requires three skinfold measurements. For men, measurement sites are the chest, abdomen and thigh; for women, they consist of the thigh, triceps and suprailiac crest, or just above the top of the hip bone. Body Fat Percentage Formula will be use as follows:
  The formula for men is: 1.10938 - (0.0008267 x the sum of the chest, abdomen and thigh measurements in millimeters) + (0.0000016 x the square of the sum of the chest, abdomen and thigh measurements in millimeters) - (0.0002574 x age) = body density
  The formula for women, also known as the Jackson-Pollock-Ward formula, is: 1.0994921 - (0.0009929 x the sum of the triceps, thigh and suprailiac measurements) + (0.0000023 x the square of the sum of the triceps, thigh and suprailiac measurements) - (0.0001392 x age) = body density

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Mutluay, Professor, Study Director — Medipol University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)